CLINICAL TRIAL: NCT07271966
Title: B6 Administration for Levetiracetam-Associated Neurobehavioral Changes and Epilepsy (BALANCE)
Brief Title: B6 Administration for Levetiracetam-Associated Neurobehavioral Changes and Epilepsy
Acronym: BALANCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00119210
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor Related Epilepsy (BTRE)
Keywords: BTRE; Vitamin B6; Levetiracetam; Katherine Peters; Pro00119210; Brain tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin B6 supplementation (Experimental)
  Interventions: Dietary Supplement: Vitamin B6 100 MG

INTERVENTIONS:
Dietary Supplement: Vitamin B6 100 MG — Patients will be prescribed 100 mg of Vitamin B6 as a supplement to take daily in the morning, by mouth for 8 to 12 weeks, in addition to the already prescribed levetiracetam.

SUMMARY:
This is a supportive care study to assess the effect of Vitamin B6 supplementation on mood-related side effects of levetiracetam in patients with brain tumors, who have already been prescribed levetiracetam for the prevention of seizures. This study will assess this effect from the perspective of both the patient and the patient's caregiver.

Patients will receive Vitamin B6 as a supplement to take daily for 8 to 12 weeks, in addition to the already prescribed levetiracetam and will undergo study assessments as well as complete self-reported questionnaires to evaluate their mood during the course of the study. Additionally, each patient will be asked to optionally identify a designated caregiver, who will complete questionnaires assessing the patient's mood changes, at the same time interval as the patient.

DETAILED DESCRIPTION:
This is a supportive care study to assess the effect of Vitamin B6 supplementation on mood-related side effects of levetiracetam in patients with brain tumors who have already been prescribed levetiracetam twice per day, for at least 6 weeks and up to 6 months for the prevention of seizures. This study will assess this effect from the perspective of both the patient and the patient's caregiver.

Patients who have been diagnosed with a primary brain tumor and who have been prescribed levetiracetam will be prescribed 100 mg of Vitamin B6 as a supplement to take daily in the morning, by mouth for 8 to 12 weeks, in addition to the already prescribed levetiracetam. Patients will undergo study assessments and will complete self-reported questionnaires to evaluate their mood at two different timepoints: one after patient enrollment and the second at the follow-up visit scheduled about 8 to 12 weeks after initiation of VitB6 supplementation .

Additionally, each patient will be asked to identify a designated caregiver, who will complete questionnaires assessing the patient's mood changes at the same time interval as the patient. A caregiver can include any person identified by the patient who is directly involved in their care and support. This includes, but is not limited to, assisting with daily living, meal preparation, transportation, medication management, financial support, coordinating health appointments, and promoting emotional well-being. The identification of a caregiver is optional and is not a requirement for patient participation.

After the patient and their caregiver complete their respective questionnaires, the study will end. Patients may choose to either continue or discontinue taking VitB6 after the study ends.

ELIGIBILITY:
Inclusion Criteria for Patients:

1. Age ≥ 18 years
2. Diagnosed with a primary brain tumor
3. Karnofsky Performance Status ≥ 70%
4. Have one or more documented seizures or transient events concerning for localization-related epilepsy requiring anti-seizure medication prophylaxis
5. Have an active immediate release levetiracetam prescription
6. Taking levetiracetam for ≥ 6 weeks and ≤ 6 months before screening
7. Baseline patient-reported mood symptoms and/or National Comprehensive Cancer Network distress thermometer score ≥ 3
8. Has access to e-mail where they can receive electronic informed consent form (ICF) and questionnaires
9. Signed ICF approved by the institutional review board (IRB)

Inclusion Criteria for Caregivers:

1. Age ≥ 18 years
2. Patient has indicated that it is acceptable to recruit their caregivers into the study
3. Able to read and write English
4. Has access to e-mail where they can receive electronic ICF and questionnaires
5. Signed ICF approved by the IRB

Exclusion Criteria for Patients:

1. Active prescription for steroids at the time of enrollment
2. Prescription for extended-release levetiracetam
3. Previous history of suicidal ideation, homicidal ideation, hallucinations, psychosis, depression leading to hospitalization, or mood disturbance leading to hospitalization
4. Prior history of alcohol use disorder or substance use disorder
5. Refractory epilepsy requiring second or third line anti-seizure medication in addition to levetiracetam at the time of enrollment
6. Patients who are currently pregnant or breastfeeding/chestfeeding
7. Patients with a pre-existing history of neuropathy
8. Known history of Vitamin B6 toxicity or deficiency
9. Prior history of gastric surgery or colectomy
10. Prior history of autoimmune disease, such as Crohn's, Ulcerative Colitis, or Celiac disease
11. Prescribed Theophylline (Aquaphyllin, Elixophyllin, Theolair, Truxophyllin) used in the treatment of asthma, chronic bronchitis, and emphysema
12. Cognitive impairment that affects the patient's ability to comprehend and provide responses to questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of VitB6 supplementation on LEV-associated mood changes in patients with BTRE, as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) anger questionnaire | From enrollment (Baseline) to follow-up at 8-12 weeks from the initiation of VitB6 supplementation
  Mean change in patient-reported PROMIS anger T-scores between baseline and the 8 to 12-week follow-up visit among patients who complete questionnaires at both timepoints. Each item on the PROMIS Anger Short Form is rated on a 5-point scale. The total score can range from 5 to 25, with higher scores indicating greater severity of anger.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, MD, PhD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No